CLINICAL TRIAL: NCT04891484
Title: Effect of Ondansetron on Spinal-induced Hypotension by Using Bupivacaine -Dexmedetomidine Mixture Intrathecally for Percutaneous Nephrolithotomy
Brief Title: Effect of Ondansetron on Spinal-induced Hypotension for Percutaneous Nephrolithotomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Mahmoud Othman, Professor of anesthesia and surgical Intensive care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS.20.09.1248
Record Dates: First submitted 2021-05-10; First posted 2021-05-18 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Percutaneous Nephrolithotomy
Keywords: Ondansetron, hypotension,vasopressor
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Two groups were enrolled in this study. They will randomized into two groups •Group S:patients will be injected with 10 ml normal saline intravenous 5 min before spinal anesthesia •Group O:patient swill be injected with 4 mg Ondansetron diluted with normal saline IV 5 minutes before spinal anesthesia
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron group (Experimental): Group O :patients will be injected with 4 mg Ondansetron diluted with normal saline IV 5 minutes before spinal anesthesia
  Interventions: Drug: Ondansetron group
- Control group (Placebo Comparator): Group S:patients will be injected with 10 ml normal saline intravenous 5 min before spinal anesthesia
  Interventions: Drug: Saline group

INTERVENTIONS:
Drug: Ondansetron group — patients will be injected with 4 mg Ondansetron diluted with normal saline IV 5 minutes before spinal anesthesia
  Arms: Ondansetron group
Drug: Saline group — patients will be injected with 10 ml normal saline intravenous 5 min before spinal anesthesia
  Arms: Control group

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is the surgical standard for treating large or complex renal stones. The stones are removed by passing a small telescope through the side of the patient directly into the kidney, so the stone can be broken up and the fragments are removed .PCNL can be performed under general anesthesia or spinal anesthesia. SA has some advantage over GA, such as lower postoperative pain, lower consumption of analgesic drugs and avoidance of side effects from multiple medications used in GA.However, SA induced sympathetic block leads to a decrease in the systemic vascular resistance and subsequent drop in the arterial blood pressure. Furthermore, anesthesia for PCNL usually requires a high sensory level reaching T4,resulting in a high incidence (nearly 33%) of hypotension. Also, to meet the long duration of surgery, drugs, ;like dexmedetomidine, are added to intrathecal local anesthetics , increasing the incidence of hemodynamic instability induced by the spinal anesthesia.

Decreasing the systemic vascular resistance (SVR) and the venous return to the heart result in a reflex vasodilation, bradycardia and hypotension. This reflex is called Bezold -Jarisch reflex and is mediated by serotonin receptors (5_HT3) located on the vagus nerve and within the wall of the cardiac ventricles.

Ondansetron; an antiemetic drug used for treatment of perioperative nausea and vomiting, was investigated as a 5HT antagonist for inhibition of Bezold - Jarisch reflex. While some studies proved its efficacy in prevention of spinal anesthesia induced hypotension , other studies could not support this conclusion .

DETAILED DESCRIPTION:
This study aims to assess the effect of Ondansetron on spinal induced hypotension when bupivacaine and dexmedetomidine are used intrathecally during spinal anesthesia for percutaneous nephrolithotomy.This prospective randomized double-blinded study will be carried out at Urology and Nephrology center, Mansoura University after approval of Institutional Research Board, Faculty of Medicine, Mansoura University. Written informed consents will be obtained from participants after explanation of the used drug and its possible consequences.

Basal readings for blood pressure, heart rate, and ECG analysis and oxygen saturation will be recorded before the start of spinal anesthesia.

Upon arrival to OR, wide bore intravenous access (20 gauge cannula) will be secured for preoperative fluid preloading (10 ml/kg ringer solution intravenously).All patients will be monitored for non-invasive blood pressure (BP), Heart rate (HR) , ECG and pulse oximetry , measurements will be recorded every 5 min for first 30 minutes then every 15 min till the end of surgery .Patients will be randomly divided into two groups, using a computer generated random table;

* Group S:patients will be injected with 10 ml normal saline intravenous 5 min before spinal anesthesia
* Group O:patients will be injected with 4mg Ondansetron diluted with normal saline IV 5 minutes before spinal anesthesia Spinal anesthesia will be delivered in the sitting position under complete aseptic condition using 25-gauge spinal needle (quinckle type), the needle will be advanced at level L 4-5 or L 3 - 4. After a clear flow of CSF, 3ml 0.5 % hyperbaric bupivacaine (15mg)will be injected followed by 5 Mcg dexmedetomidine in insulin syringe diluted to 1ml .After anesthesia, patients will be positioned supine immediately, sensory level will be assessed each 2 minutes by pinprick test, a sensory block at T4-6 will be considered sufficient to start surgery.o BP, HR and oxygen saturation will be recorded every 5 minutes for first 30 minutes then every 15 minutes till the end of surgery. Hypotension will be defined as a decrease blood pressure more than 20% of basal BP or decrease systolic than 90 mmHg and will be treated with IV ephedrine (5mg bolus). Bradycardia will be defined as heart rate less than 50 beat / min and will be treated with IV atropine (0.5mg).The maximum level of sensory block will be assessed every 2 minutes till reaching maximum level of sensory block by pin prick test or cold sensation using alcohol swab.The incidence of ECG changes(dysrhythmia, ST changes).The incidence of pruritus.The incidence of nausea and /or vomiting.Postoperative data( HR, BP, SPo2) will be measured every 15 minutes for 2 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for PCNL surgery.
2. ASA classification I or II

Exclusion Criteria:

1. Patient refusal
2. Contraindication to spinal anesthesia.
3. Known allergy to Ondansetron.
4. Uncontrolled hypertensive patient.
5. Ischemic heart diseases.
6. Moderate to severe stenotic valve lesion.
7. Atrial fibrillation.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
The incidence of hypotension during spinal anesthesia for percutaneous nephrolithotomy | perioperative time for two hours postoperatively
  The incidence of hypotension with mean pressure below 60 mmhg during spinal anesthesia for PCNL

SECONDARY OUTCOMES:
The severity of hypotension | perioperative time for two hours postoperatively
  The severity of hypotension with mean blood pressurer either mild (less than 60 mmHg), or moderate(less than50 mmHg or severe (less than 40mmHg)
The duration and number of hypotension episodes | perioperative time for two hours postoperatively
  The duration of each hypotension episode
The need of vasopressors (ephedrine and noradrenaline) . | perioperative time for two hours postoperatively
  The need and the dose of vasopressors (ephedrine and noradrenaline) .
The incidence of bradycardia Intraoperative | perioperative time for two hours postoperatively
  The incidence of bradycardia Intraoperative
The incidence of perioperative nausea and vomiting | perioperative time for two hours postoperatively
  The incidence of perioperative nausea and vomiting
The incidence of perioperative shivering | perioperative time for two hours postoperatively
  The incidence of perioperative shivering
The incidence of perioperative pruritus | perioperative time for two hours postoperatively
  The incidence of perioperative pruritus

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Othman, MD, Principal Investigator — Department of anesthesia ,Urology and nephrology center ,Faculty of medicine,Mansoura university
Locations (1):
- Urology and nephrology center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No